CLINICAL TRIAL: NCT02691663
Title: Dietary Acid Load, Kidney Function and Disability in Elderly
Acronym: BICARB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00034474; R21AG051866 (NIH)
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Results first posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-06

CONDITIONS: Chronic Kidney Disease; Disability
Keywords: Geriatric; bicarbonate
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral bicarbonate supplementation group (Active Comparator): 0.3 meq/kg/day NaHCO3 capsules
  Interventions: Dietary Supplement: Oral bicarbonate supplementation
- Placebo group (Placebo Comparator): Methylcellulose capsules
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oral bicarbonate supplementation
  Arms: Oral bicarbonate supplementation group
Dietary Supplement: Placebo
  Arms: Placebo group

SUMMARY:
The purpose of this research study is to determine the effect of a bicarbonate supplement on kidney function and physical function.

DETAILED DESCRIPTION:
Physical decline and frailty result from age- and disease-related impairments in organs and tissues. Frailty research has focused on the musculoskeletal, neurological and circulatory systems; yet interventions targeting these systems had limited success in preventing and treating functional decline. Given the aging of the US population, additional avenues for intervention development are urgently needed. Fragility and disability in people ≥65 strongly correlate with declining kidney function and are evident even in early stages of chronic kidney disease (CKD). Moreover, CKD is highly prevalent in the elderly and associates with sarcopenia, osteopenia, and increased incidence of fractures/falls with hospitalization. Low serum bicarbonate and impaired acid-base homeostasis, also common in CKD, are increasingly appreciated as contributors to functional decline with advancing age. With aging, the adaptive response of the kidney to low serum bicarbonate and high metabolic acid load becomes maladaptive, facilitating CKD progression. Conversely, in adult patients with CKD, maintenance of serum bicarbonate at 24 meq/L with oral bicarbonate supplementation or increased consumption of base-forming foods slows CKD progression.

The study investigators propose the current study and protocol based on the evidence summarized above and our preliminary studies, which suggest that: In the Health Aging and Body Composition cohort (age 70-79) lower dietary acid load associates with stable kidney function over a 7-year follow-up, independent of age, race, gender, BMI, diabetes, hypertension or smoking status; metabolomics analysis in participants of the African American Diabetes Heart Study suggested that it is feasible to segregate a urine metabolomics profile in the early stages of CKD (stages 2 and 3), and that lower consumption of base-forming fruits and vegetables and higher rates of acid excretion may be associated with CKD and its progression.

The investigators therefore hypothesized that decreasing metabolic acid production by titrating dietary acid load may ameliorate the generally expected, age-related decline in kidney function, decrease loss of lean body mass, preserve physical function, and ameliorate disability. This is not a treatment study as the investigators are exploring the effects of bicarbonate on these age-related issues.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 +years of age
* Short physical performance battery (SPPB) score>3
* Estimated glomerular filtration rate (eGFR) 30-89
* Net endogenous acid production (NEAP) >=40 mEq/d
* Willing to provide informed consent and agrees to randomization
* Not involved in another intervention study

Exclusion Criteria:

* Uncontrolled (>160 mg/dl fasting blood glucose), insulin-dependent diabetes and/or uncontrolled hypertension (Systolic Blood Pressure >160, Diastolic BP>100)
* a current diagnosis of psychotic disorder
* take more than 14 alcoholic drinks per week
* plan to relocate out of the study area within the next year
* self-reported inability to walk across a room
* those who reside in nursing homes
* have difficulty communicating with study personnel due to speech or language or hearing problems
* had cancer requiring treatment in the past 1 year
* lung disease requiring regular use of corticosteroids or of supplemental oxygen
* cardiovascular disease (Class III or IV congestive heart failure)
* significant valvular disease, uncontrolled angina
* myocardial infarction, major heart surgery (i.e., valve replacement or bypass surgery) in past 6 months
* stroke, deep vein thrombosis, or pulmonary embolus in the past 6 months, Parkinson's disease or other progressive neurological disorder
* other medical or behavioral factors that in the judgment of the principal investigator may interfere with study participation or the ability to follow the intervention
* clinical judgment concerning safety or noncompliance
* Individuals with BMI <18.5; or weight loss >4% in last 6 months
* Montreal Cognitive Assessment (MoCA) score under 24
* End Stage Renal Disease (ESRD) on dialysis or primary kidney disease
* Other illness of such severity that life expectancy is less than 12 months
* Smoking; defined as not smoking for more than a year prior to the study
* Serum Bicarbonate (HCO3)>30 milliequivalents per liter (mEq/L); serum potassium out of normal range

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 196 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Snezana Petrovic, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 196 subjects signed consent; all except 83 were screen failures; 83 subjects were randomized
Groups:
- Oral Bicarbonate Supplementation Group: 0.3 meq/kg/day NaHCO3 capsules
  Oral bicarbonate supplementation
- Placebo Group: Methylcellulose capsules
  Placebo
Period: Overall Study
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Started | 41 | 42
Completed | 33 | 35
Not Completed | 8 | 7
Not completed — Screen failure after baseline | 2 | 2
Not completed — withdrawn after Follow up 1 visit | 2 | 2
Not completed — Withdrawn after Follow up 2 | 1 | 1
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group | Total
Number analyzed (Participants) | 41 | 42 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.3 (5.9) | 72.3 (5.5) | 72.8 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 49
  Male | 17 | 17 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 40 | 41 | 81
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 36 | 37 | 73
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Blood Bicarbonate
Description: measurement taken from a blood sample; measures how much carbon dioxide is in your blood; a normal result is between 23 and 29 millimoles per liter (mmol/L) for adults
Time Frame: baseline
Population: PI is reporting blood bicarbonate from blood gas measurement as a surrogate of NEA because a percentage of NEA samples could not be accurately measured due to technical issues.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 41 | 42
mmol/L | 22.8 (2.3) | 23.2 (2.4)

2. Primary Outcome: Blood Bicarbonate
Description: as for outcome 1
Time Frame: six months post baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 33 | 35
mmol/L | 23.8 (2.3) | 23.3 (2.1)

3. Secondary Outcome: Percentage of Screened Participants Randomized
Description: The number of participants randomized divided by the number of participants screened. Count of participants reflects the number of participants randomized.
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study: This includes all participants in the study, including participants screened and enrolled.
Arm/Group | Overall Study
Number analyzed (Participants) | 196
Participants | 83

4. Secondary Outcome: Percent Adherence: Percentage of Pills Taken
Description: based on pill count
Time Frame: 6 months post baseline
Measure: Mean (Standard Deviation); unit: percentage of pills
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 34 | 37
percentage of pills | 90.5 (12.9) | 85.2 (21.4)

5. Secondary Outcome: Carbon Dioxide Blood Test
Description: Blood test that measures the total dissolved Carbon dioxide in blood; expressed in milliequivalents per liter (mEq/L)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 41 | 42
mEq/L | 35.4 (3.6) | 36.5 (4.1)

6. Secondary Outcome: Carbon Dioxide Blood Test
Description: Blood test that measures the total dissolved Carbon dioxide in blood; expressed in milliequivalents per liter (mEq/L)
Time Frame: six months post baseline
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 33 | 35
mEq/L | 36.9 (3.9) | 37.0 (3.5)

7. Secondary Outcome: 400 Meter Walk Time
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 41 | 42
minutes | 6.3 (1.2) | 6.3 (1.4)

8. Secondary Outcome: 400 Meter Walk Time
Time Frame: three months post baseline
Population: 1 bicarb Participant refused 400m walk at the 3-month visit.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 33 | 37
minutes | 6.3 (1.0) | 6.5 (1.7)

9. Secondary Outcome: 400 Meter Walk Time
Time Frame: six months post baseline
Population: 3 participants (2 bicarb and 1 placebo) refused 400m walk at the 6-month visit
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 31 | 34
minutes | 6.1 (1.0) | 6.3 (1.5)

10. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR)
Description: a measurement from a blood sample; shows how well kidneys are working According to the National Institutes of Health (NIH), normal results range from 60 to 120 mL/min/1.73 m2. Older people will have lower than normal eGFR levels, because eGFR decreases with age
Time Frame: baseline
Population: creatinine and MDRD equation
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 41 | 42
mL/min/1.73m^2 | 65.4 (13.1) | 66.9 (15.1)

11. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR)
Description: as for outcome 10
Time Frame: three months post baseline
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 34 | 37
mL/min/1.73m^2 | 66 (15.3) | 63.9 (15.7)

12. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR)
Description: as for outcome 10
Time Frame: six months post baseline
Population: creatinine and MDRD equation
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 33 | 35
mL/min/1.73m^2 | 64.7 (16.0) | 64.7 (17.8)

13. Secondary Outcome: Measurement of Kidney Function (eGFR) at Baseline.
Description: as for outcome 10
Time Frame: baseline
Population: cystatin C and CKD Epi equation
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 41 | 42
mL/min/1.73m^2 | 81.3 (19.1) | 81.3 (21.0)

14. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR) - Measurement of Kidney Function After 6 Months Post Baseline
Description: as for outcome 10
Time Frame: six months post baseline
Population: cystatin C and CKD Epi equation
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 33 | 35
mL/min/1.73m^2 | 80.1 (20.3) | 81.0 (20.4)

15. Secondary Outcome: Hip Bone Mineral Density
Description: Bone Mineral Density tests can identify osteoporosis, determine the risk for fractures (broken bones), and measure the response to osteoporosis treatment.
Time Frame: baseline
Population: No baseline dual energy x-ray absorptiometry (DXA) scans were completed for 3 bicarb and 1 placebo participants.
Measure: Mean (Standard Deviation); unit: g/cm^3
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 38 | 41
g/cm^3 | .94 (.15) | .93 (.18)

16. Secondary Outcome: Hip Bone Mineral Density
Description: as for outcome 15
Time Frame: six months post baseline
Population: No 6-month DXA scans were completed for 1 bicarb and 3 placebo participants.
Measure: Mean (Standard Deviation); unit: g/cm^3
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 32 | 32
g/cm^3 | .93 (.15) | .91 (.15)

17. Secondary Outcome: Femoral Neck Bone Mineral Density
Description: as for outcome 15
Time Frame: baseline
Population: No baseline DXA scans were completed for 3 bicarb and 1 placebo participants.
Measure: Mean (Standard Deviation); unit: g/cm^3
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 38 | 41
g/cm^3 | .76 (.13) | .74 (.15)

18. Secondary Outcome: Femoral Neck Bone Mineral Density
Description: as for outcome 15
Time Frame: six months post baseline
Population: No 6-month DXA scans were completed for 1 bicarb and 3 placebo participants.
Measure: Mean (Standard Deviation); unit: g/cm^3
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 32 | 32
g/cm^3 | .74 (.13) | .72 (.14)

19. Secondary Outcome: Average Body Mass Index (BMI)
Time Frame: baseline
Population: baseline BMI is missing for 4 participants (3 bicarb and 1 placebo) due to missing height measurement (height was only measured at the screening visit).
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 38 | 41
kg/m^2 | 27.6 (5.3) | 28.1 (4.8)

20. Secondary Outcome: Average Body Mass Index (BMI)
Time Frame: three months post baseline
Population: 3-month BMI is missing for 4 participants (3 bicarb and 1 placebo) due to missing height measurement (height was only measured at the screening visit).
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 31 | 36
kg/m^2 | 26.6 (4.4) | 28.3 (4.9)

21. Secondary Outcome: Average Body Mass Index (BMI)
Time Frame: six months post baseline
Population: 6-month BMI is missing for 4 participants (3 bicarb and 1 placebo) due to missing height measurement (height was only measured at the screening visit).
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 30 | 34
kg/m^2 | 26.3 (4.4) | 28.1 (4.9)

22. Secondary Outcome: Urinary Albumin to Creatinine Ratio (ACR)
Description: The albumin-to-creatinine ratio (ACR) is the first method of preference to detect elevated protein, measuring urinary ACR in a spot urine sample. ACR is calculated by dividing albumin concentration in milligrams by creatinine concentration in grams.
Time Frame: baseline
Population: baseline ACR is missing for 7 participants (3 bicarb and 4 placebo).
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 38 | 38
mg/g | 25.1 (23.2) | 53.8 (139.7)

23. Secondary Outcome: Urinary Albumin to Creatinine Ratio (ACR)
Description: as for outcome 22
Time Frame: three months post baseline
Population: 3-month ACR is missing for 10 participants (5 bicarb and 5 placebo).
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 29 | 32
mg/g | 33.9 (40.3) | 52.8 (126.0)

24. Secondary Outcome: Urinary Albumin to Creatinine Ratio (ACR)
Description: as for outcome 22
Time Frame: six months post baseline
Population: 6-month ACR is missing for 5 participants (0 bicarb and 5 placebo).
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 33 | 30
mg/g | 45.1 (119.8) | 80.4 (254.7)

25. Other Pre Specified Outcome: Net Endogenous Acid Production (NEAP)
Description: (mEq/day) by the kidney
Time Frame: 6 months post randomization
Population: 6 month data missing for one subject in bicarbonate (bicarb) arm
Measure: Mean (Standard Deviation); unit: mEq/day
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 32 | 35
mEq/day | 75.0 (37.6) | 73.8 (39.0)

26. Other Pre Specified Outcome: Net Endogenous Acid Production (NEAP)
Description: mEq/day by the kidney
Time Frame: 3 months post randomization
Measure: Mean (Standard Deviation); unit: mEq/day
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 34 | 37
mEq/day | 79.4 (33.2) | 75.3 (38.7)

27. Other Pre Specified Outcome: Net Endogenous Acid Production (NEAP)
Description: mEq/day by the kidney
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mEq/day
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
Number analyzed (Participants) | 33 | 35
mEq/day | 79.3 (29.7) | 72.1 (23.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected after subjects signed consent until the end of subject participation over a period of 6 months.
Arm/Group | Oral Bicarbonate Supplementation Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/42
Serious Adverse Events (participants affected / at risk) | 1/41 | 1/42
Other Adverse Events (participants affected / at risk) | 8/41 | 8/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Bicarbonate Supplementation Group (N=41) | Placebo Group (N=42)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Transient Ischemic Attack (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Bicarbonate Supplementation Group (N=41) | Placebo Group (N=42)
indigestion (Gastrointestinal disorders) | 1 (1) | 2 (2)
Elevated Blood Pressure (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
edema (Cardiac disorders) | 2 (2) | 1 (1)
atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Broken fifth toe right side (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT02691663/Prot_SAP_000.pdf